CLINICAL TRIAL: NCT03065608
Title: Evaluation of C-reactive Protein Level in the Group of Patient With Pain Form of Temporomandibular Joint Dysfunction
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Malgorzata Pihut, Associate Professor, Jagiellonian University
Other Study IDs: KBET/125/L/2013
Record Dates: First submitted 2017-02-17; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The study group included 36 patients with pain form of dysfunction.
- Control Group: The control group consisted of 36 patients with painless form of disorder.

SUMMARY:
Temporomandibular joints dysfunction is a functional disorder concern with the abnormal functioning of the muscles of the stomatognathic system, temporomandibular joints involved in the dynamic movements of the jaw and surrounding structures.

The aim of the study was to compare the level of C-reactive protein in patients with pain and painless form of temporomandibular joints dysfunction.

DETAILED DESCRIPTION:
Temporomandibular joints dysfunction is a functional disorder concern with the abnormal functioning of the muscles of the stomatognathic system, temporomandibular joints involved in the dynamic movements of the jaw and surrounding structures.

The aim of the study was to compare the level of C-reactive protein in patients with pain and painless form of temporomandibular joints dysfunction.

Material and methods The research material consisted of 72 patients who reported to the prosthetic treatment because of temporomandibular joint dysfunction. The study group included 36 patients with pain form of dysfunction, and control group - 36 patients with painless form of disorder. Each patient underwent specialized examination of functional disorders, in order to diagnose the type of dysfunction and commissioned to carry out a study of the blood test concern with evaluation of the C-reactive protein (CRP) level in the same analytical laboratory.

The results of the investigation were subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Factors of inclusion in the study are: pain form of temporomandibular joints dysfunction, the required age range, a good general state of health (particularly with regard to cardiac and metabolic disorders).

Exclusion Criteria:

* Factors for exclusion from the research include: the will of the patient, the emergence of general diseases, trauma, or local inflammation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled a group of 72 patients, aged 21 to 48 years, of both sexes, who reported to the prosthodontic treatment in Consulting Room of Temporomandibular Joint Dysfunction at Dental Institute at Jagiellonian University in Cracow, between January 2015 to February 2017, due to the pain and painless form of the temporomandibular joints dysfunction, and acoustic symptoms, accompanied by excessive tension of masticatory muscle. Symptoms persisted from 3 to 12 months prior to beginning of the treatment.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
By means of the CRP-level it will be verified if the temporomandibular joint dysfunctions are associated with inflammations of the temporomandibular joints. | 12 months
  The aim of the study is to avaluation of the level of C-reactive protein in patients treated prosthetically due to the pain form of temporomandibular joints dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Pihut, Associate Professor, Principal Investigator — Jagiellonian University; Piotr Ceranowicz, MD,PhD,, Study Chair — Jagiellonian University; Andrzej Gala, DDS,PhD,, Study Chair — Jagiellonian University; Mieszko Więckiewicz, DMD,PhD,, Study Chair — Wroclaw Medical University

IPD SHARING:
Plan to Share IPD: No